CLINICAL TRIAL: NCT06265727
Title: A Phase 1/2 Study to Investigate the Safety, Pharmacokinetics, and Efficacy of CRB-701, an Antibody-drug Conjugate Targeting Nectin-4, in Patients With Advanced Solid Tumors
Brief Title: A Phase 1/2 Study to Investigate CRB-701 in Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Corbus Pharmaceuticals Inc. (Industry)
Collaborators: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRB-701-01
Record Dates: First submitted 2024-02-08; First posted 2024-02-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor, Adult
Keywords: nectin-4
MeSH Terms: interventions — spartalizumab

STUDY DESIGN:
Intervention Model Description: A three part study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Part A Dose Escalation - CRB-701 Dose Level 1 (Experimental): CRB-701 Dose level 1, intravenous infusion over 30 mins, Dose schedule 1
  Interventions: Drug: CRB-701
- Part A Dose Escalation - CRB-701 Dose Level 2 (Experimental): CRB-701 Dose Level 2, intravenous infusion over 30 mins, Dose schedule 1
  Interventions: Drug: CRB-701
- Part A Dose Escalation - CRB-701 Dose Level 3 (Experimental): CRB-701 Dose Level 3, intravenous infusion over 30 mins, dose schedule 1
  Interventions: Drug: CRB-701
- Part A Dose Escalation - CRB-701 Dose Level 4 (Experimental): CRB-701 Dose Level 4, intravenous infusion over 30 mins, dose schedule 1
  Interventions: Drug: CRB-701
- Part B Dose Optimization: CRB-701 High dose (Experimental): Selected high dose of CRB-701, intravenous infusion over 30 mins, dose schedule 1
  Interventions: Drug: CRB-701
- Part B Dose Optimization: CRB-701 low dose (Experimental): Selected Low dose of CRB-701, intravenous infusion over 30 mins
  Interventions: Drug: CRB-701
- Part C Dose Expansion - Cohort 1 (Experimental): Recommended CRB-701 dose and schedule, intravenous infusion over 30 mins followed by infusion with anti-PD-1
  Interventions: Drug: CRB-701; Drug: Anti-PD-1
- Part C Dose Expansion - Cohort 2 (Experimental): Recommended CRB-701 dose and schedule, intravenous infusion over 30 mins
  Interventions: Drug: CRB-701
- Part C Dose Expansion - Cohort 3 (Experimental): Recommended CRB-701 dose and schedule, intravenous infusion over 30 mins followed by infusion with anti-PD-1
  Interventions: Drug: CRB-701; Drug: Anti-PD-1
- Part C Dose Expansion - Cohort 4 (Experimental): Recommended CRB-701 dose and schedule, intravenous infusion over 30 mins
  Interventions: Drug: CRB-701
- Part C Dose Expansion - Cohort 5 (Experimental): Recommended CRB-701 dose and schedule, intravenous infusion over 30 mins followed by infusion with anti-PD-1
  Interventions: Drug: CRB-701; Drug: Anti-PD-1
- Part B Dose Optimization: CRB-701 high dose combined with anti-PD-1 (Experimental): Selected high dose of CRB-701, intravenous infusion over 30 mins followed by infusion with anti-PD-1
  Interventions: Drug: CRB-701; Drug: Anti-PD-1
- Part B Dose Optimization: CRB-701 low dose combined with anti-PD-1 (Experimental): Selected low dose of CRB-701, intravenous infusion over 30 mins followed by infusion with anti-PD-1
  Interventions: Drug: CRB-701; Drug: Anti-PD-1
- Part C Dose Expansion - Cohort 6 (Experimental): Recommended CRB-701 dose and schedule, intravenous infusion over 30 mins
  Interventions: Drug: CRB-701
- Part C Dose Expansion - Cohort 7 (Experimental): Recommended CRB-701 dose and schedule, intravenous infusion over 30 mins followed by infusion with anti-PD-1
  Interventions: Drug: CRB-701; Drug: Anti-PD-1

INTERVENTIONS:
Drug: CRB-701 — Nectin-4 targeted Antibody Drug Conjugate (ADC)
Drug: Anti-PD-1 — checkpoint inhibitor
  Arms: Part B Dose Optimization: CRB-701 high dose combined with anti-PD-1; Part B Dose Optimization: CRB-701 low dose combined with anti-PD-1; Part C Dose Expansion - Cohort 1; Part C Dose Expansion - Cohort 3; Part C Dose Expansion - Cohort 5; Part C Dose Expansion - Cohort 7

SUMMARY:
The goal of this clinical trial is to define a safe and effective dose of CRB-701 for participants with solid tumors that are expressing a protein called nectin-4.

The main questions it aims to answer are:

What is the the safe and effective dose of CRB-701? What cancers can be treated effectively with CRB-701?

Participants will be asked to attend clinic and be given a intravenous infusion of CRB-701. They will have blood tests, CT or MRI Scans, and other assessments to measure whether CRB-701 has an effect on tumors.

DETAILED DESCRIPTION:
This is a three-part open-label, Phase 1/2 clinical trial designed to evaluate the safety, PK, and efficacy of CRB-701 in participants with advanced solid tumors expressing nectin-4.

Part A will include solid tumor types known to express nectin-4. Dose escalation will be guided by the Bayesian optimal interval (BOIN) design to determine the Maximum Tolerated Dose (MTD) of CRB-701. Four (4) dose groups are pre-determined. Dose escalation/de-escalation decisions are made based on the occurrence of DLT.

Part B will evaluate two dose levels of CRB-701 alone and in combination with anti-PD-1 by using a time-to-event Bayesian optimal Phase 2 study design to optimize the dose of CRB-701 in one or more separate cohorts of participants with nectin-4-positive tumors.

During Part C, the recommended dose level of CRB-701 for further exploration defined in Part B will explore CRB-701 alone or combined with anti-PD-1 in up to seven separate cohorts of participants with advanced tumors known to express Nectin-4.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of select advanced or metastatic nectin-4 expressing solid tumors that have progressed having exhausted all appropriate lines of therapy or have no other standard therapy with proven clinical benefit. In Part C, HNSCC participants may enroll as first-line therapy.

Exclusion Criteria:

* Active of uncontrolled CNS metastases
* History of solid tumors other than the diseases under study
* History of and/or current cardiovascular events or conditions in the previous 6 months
* Pre-existing >/= Grade 2 neuropathy
* Hemoglobin A1C (HbA1C) >/= 8%, uncontrolled diabetes mellitus or know diabetic neuropathy
* Active ocular disease at baseline
* Chronic severe liver disease or live cirrhosis
* Interstitial lung disease or pneumonitis within 6 months on initiating treatment on study
* Other significant cormorbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-01-16 (Estimated); Study Completion 2027-01-27 (Estimated)

PRIMARY OUTCOMES:
Part A: To confirm the safety and tolerability and determine MTD and PADR for CRB-701 | 21 days
  Occurrence of Dose Limiting Toxicities as defined in the protocol
Part B & C: To evaluate efficacy in terms of Objective Response Rate (ORR) | Up to 6 months
  ORR is the percentage of participants that achieve a response (CR + PR) using RECIST 1.1

SECONDARY OUTCOMES:
Parts A, B, & C: To characterize the safety profile of CRB-701 | Up to 6 months
  Numbers of treatment emergent adverse events with severity determined using NCI CTCAE v5.0 after single or multiple doses of CRB-701 or single and multiple doses of CRB-701 and an anti-PD-(L)1 therapy
Maximum observed plasma concentration of CRB-701 [total ADC] (Cmax) | Approximately 9 weeks
  Maximum observed plasma concentration of total ADC after single and multiple doses
Maximum observed plasma concentration of free MMAE (Cmax) | Approximately 9 weeks
  Maximum observed plasma concentration of free MMAE after single and multiple doses
Part B & C : To evaluate efficacy in terms of Disease Control Rate (DCR) | Up to 6 months
  DCR is the sum of percentage of participants meeting the definition of Complete Response (CR), Partial Response (PR) or Stable Disease (SD) for at least 4 months using RECIST 1.1
Maximum observed plasma concentration of Total CRB-701 antibody [Tab] (Cmax) | Approximately 9 weeks
  Maximum observed plasma concentration of free MMAE after single and multiple doses
Time to reach Cmax of Total CRB-701 [Total ADC] (Tmax) | Approximately 9 weeks
  The amount of time to reach Cmax after single and multiple dose administration of CRB-701 (Total ADC)
Time to reach Cmax of free MMAE (Tmax) | Approximately 9 weeks
  The amount of time to reach Cmax after single and multiple dose administration of free MMAE
Time to reach Cmax of Total CRB-701 antibody [Tab] (Tmax) | Approximately 9 weeks
  The amount of time to reach Cmax after single and multiple dose administration of Tab
Time to reach Cmax of Total CRB-701 antibody [Tab] (Cmax) | Approximately 9 weeks
  Maximum observed plasma concentration of free MMAE after single and multiple doses
Total Area Under the plasma concentration-time curve of Total CRB-701 [total ADC] (AUC) | Approximately 9 weeks
  Maximum observed plasma concentration of free MMAE after single and multiple doses
Total Area Under the plasma concentration-time curve of free MMAE (AUC) | Approximately 9 weeks
  Area under the plasma concentration versus time curve after single and multiple dose administration of free MMAE
Total Area Under the plasma concentration-time curve of Total CRB-701 antibody [Tab] (AUC) | Approximately 9 weeks
  Area under the plasma concentration versus time curve after single and multiple dose administration of Tab

CONTACTS AND LOCATIONS:
Overall Officials: David Pinato, MD, Principal Investigator — Imperial College London; Ian Hodgson, PhD, Study Director — Corbus International Ltd; Ari Rosenberg, MD, Principal Investigator — University of Chicago
Locations (41):
- United States (15):
  - O'Neal Comprehensive Cancer Center at University of Alabama-Birmingham, Birmingham, Alabama
  - City of Hope Cancer Center, Duarte, California
  - Moores Cancer Centre at UC San Diego Health, San Diego, California
  - Helen Diller Family Comprehensive Cancer Center - UCSF, San Francisco, California
  - Rocky Mountain Cancer Centres, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - Hope and Healing Cancer Center, Hinsdale, Illinois
  - Dana-Faber Cancer Institute, Boston, Massachusetts
  - Nebraska Hematology Oncology, Lincoln, Nebraska
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Texas Oncology, Tyler, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Fred Hutchinson Cancer Center at University of Washington, Seattle, Washington
- France (4):
  - ICM-Val d'Aurelle, Montpellier
  - CHU de Poitiers, Poitiers
  - Institut de Cancerologie de l'Ouest, Saint-Herblain
  - Gustave Roussy, Villejuif
- Italy (4):
  - Careggi University Hospital, Florence
  - European Institute of Oncology IRCCS, Milan
  - Fondazione Policlinico Gemelli, IRCCS, Rome
  - Centro Richerche Cliniche di Verona, Verona
- Institute of Oncology/ARENSIA Exploratory Medicine, Chisinau, Moldova
- Romania (4):
  - Aresnsia Research Clinic Bucharest, Bucharest
  - Aresnsia Research Clinic Cluj-Napoca, Cluj-Napoca
  - Centrul de Oncologie Sf. Nectarie, Iași
  - Centrul de Oncologie Euroclinic, Iași
- Spain (4):
  - Barcelona IOB Hospital Quironsalud (NEXT), Barcelona
  - Vall d-Hebron Institut d'Oncologia, Barcelona
  - Fundacion Jimenez Diaz (START), Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (9):
  - University of Birmingham NHS Foundation Trust, Birmingham
  - University of Cambridge NHS Foundation Trust, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Leeds University Hospitals NHS Trust, Leeds
  - Guy's and St Thomas' Clinical Research Facility, London
  - Imperial Experimental Cancer Medicine Centre, London
  - The Christie Hospital, Manchester
  - University of Liverpool - Clatterbridge Medical Centre, Metropolitan Borough of Wirral
  - University of Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No